CLINICAL TRIAL: NCT04268368
Title: Incidence, Clinical Management and Molecular Factors Associated With the Development of Immune-related Adverse Events in Cancer Patients Receiving PD-1 and PD-L1 Inhibitors: a Prospective Observational Study
Brief Title: Immune Related-adverse Events in Patients Receiving Immune Checkpoint Inhibitors
Acronym: ICI-DISCOVER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Armando Gabrielli, Full Professor, Università Politecnica delle Marche
Other Study IDs: ICI-DISCOVER
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cancer; Lung Cancer; Renal Cell Carcinoma; Melanoma
Keywords: cancer; immune checkpoint inhibitors; immune related adverse events; nivolumab; pembrolizumab; avelumab; durvalumab; atezolizumab
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Carcinoma, Renal Cell; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected for the preparation of serum and plasma at the baseline visit and at follow-up visits for all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The recent introduction of anti-PD-1 (nivolumab and pembrolizumab) and anti- PD-L1 (atezolizumab, durvalumab, avelumab) immune checkpoint inhibitors revolutionized oncological guidelines. Durable responses and prolongation of survival with these agents come at the price of the development of immune related adverse events (irAEs). Innovative tools are required in order to manage irAEs and to prevent their potential relapse, with the goal to improve the outcome of patients. In this regard, the Investigators aim to develop a multidisciplinary clinical pathway for cancer patients that are treated with immune checkpoint inhibitors.

DETAILED DESCRIPTION:
Recent evidences in immuno-oncology showed an important role of the immune system in tumor control. In fact, immune response, both innate and adaptive one, is the first defensive mechanism against cancer. However, several tumors, during their progression, develop an immune-tolerance characterized by the activation of immune inhibitory pathways including PD-1 and PD-L1.

The recent introduction of anti-PD-1 (nivolumab and pembrolizumab) and anti-PD-L1 (atezolizumab, durvalumab, avelumab) immune checkpoint inhibitors revolutionized oncological guidelines.

Currently, the aforementioned agents are approved for the treatment of advanced malignant melanoma; non-small cell lung cancer (NSCLC) and renal cell carcinoma (RCC) and the number of treatment indications for immune checkpoint inhibitors is expanding. Durable responses and prolongation of survival with these agents come at the price of the development of immune-related adverse events (irAEs).

Immune-related adverse events are due to the loss of immune-tolerance towards structures of the self, with the induction of chronic inflammation with an autoimmune mechanism that can involve numerous organs and systems. The most frequent irAEs reported in clinical trials are represented by skin toxicity, gastrointestinal toxicity, endocrine toxicity, pulmonary toxicity, and others such as polymyalgia rheumatica, polyarthritis, myositis, nephritis, polyradiculoneuritis, encephalitis and myocarditis.

The irAEs reported in clinical trials with nivolumab amount to a maximum of 85% considering all grade of toxicities, while approximately 75% of patients treated with pembrolizumab presented irAEs. Grade 3/4 irAEs were reported in 10% of patients treated with anti-PD-1. With atezolizumab fewer patients had treatment-related grade 3 or 4 adverse events (15%).

In most cases, irAEs occur within some weeks after starting of immunotherapy; however these toxicities have been reported later and also years after treatment discontinuation. The development of irAEs is associated with significant morbidity and mortality in cancer patients treated with immune checkpoint inhibitors, and therefore they may significantly affect the quality of life, even in patients achieve the control of neoplastic disease.

The overseeing, early diagnosis and clinical management of immune checkpoint inhibitors' toxicities in the clinical setting are, currently, not standardized.

Innovative tools are required in order to manage irAEs and to prevent their potential relapse, with the goal to improve the outcome and quality of life of these patients.

In this regard, the Investigators also aim to evaluate a model of multidisciplinary clinical pathway for cancer patients that are treated with immune checkpoint inhibitors in order to improve their management and also ameliorate the quality of life of patients that develop irAEs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients above 18 years of age;
2. Cyto-histological diagnosis of one of the following cancers:

   1. advanced melanoma;
   2. metastatic or locally advanced non-small cell lung cancer;
   3. advanced renal cell carcinoma;
   4. metastatic or locally advanced urotelial carcinoma;
   5. squamous cell carcinoma of the head and neck;
   6. Hodgkin lymphoma;
   7. Merkel-cell carcinoma;
3. New prescription of one of the following PD-1/PD-L1 inhibitors:

   1. nivolumab
   2. pembrolizumab
   3. atezolizumab
   4. avelumab
   5. durvalumab alone or in combination therapy, following the indications of the Italian regulatory agency (AIFA).

Exclusion Criteria:

1. Patients that refuse and/or are not able to sign the Informed Consent;
2. Parents/guardians or subjects who, in the opinion of the Investigator, may be noncompliant with study schedules or procedures;
3. No contraindications to the treatment with PD-1/PD-L1 antibodies, following the indications of the Italian regulatory agency (AIFA).

Subjects that do not meet all of the enrollment criteria may not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referring to the Oncology and Hematology Clinics of the Azienda Ospedaliero- Universitaria Ospedali Riuniti di Ancona (Italy) may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of irAEs | 24 months
  To determine the incidence and the characteristics of irAEs in a real-world setting
Risk factors for irAEs | 24 months
  To determine the risk factors for the development of irAEs
Impact of irAEs | 24 months
  To determine the impact of irAEs on patients' prognosis
Therapies of irAEs | 24 months
  To determine the effect of immunosuppressive therapies on tumor progression and patient's prognosis

SECONDARY OUTCOMES:
Clinical care pathway | 24 months
  To set up an integrated clinical care pathway for cancer patients that developed an irAE following immune checkpoint inhibitor administration
Quality of life | 24 months
  The quality of life will be measured by means of the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30). It is composed by five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Biomarkers | 24 months
  To evaluate potential biomarkers that may predict the development of irAEs and/or the response to treatment in biological samples from cancer patients treated with immune checkpoint inhibitors
Exploratory analyses | 24 months
  To get better insights on the biological basis of irAEs the response to treatment in biological samples from cancer patients treated with immune checkpoint inhibitors

CONTACTS AND LOCATIONS:
Locations (1):
- Università Politecnica delle Marche, Ancona, AN, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brahmer JR, Lacchetti C, Schneider BJ, Atkins MB, Brassil KJ, Caterino JM, Chau I, Ernstoff MS, Gardner JM, Ginex P, Hallmeyer S, Holter Chakrabarty J, Leighl NB, Mammen JS, McDermott DF, Naing A, Nastoupil LJ, Phillips T, Porter LD, Puzanov I, Reichner CA, Santomasso BD, Seigel C, Spira A, Suarez-Almazor ME, Wang Y, Weber JS, Wolchok JD, Thompson JA; National Comprehensive Cancer Network. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2018 Jun 10;36(17):1714-1768. doi: 10.1200/JCO.2017.77.6385. Epub 2018 Feb 14. PMID 29442540